CLINICAL TRIAL: NCT05526599
Title: The Association of Marital Status With Kidney Cancer Surgery Morbidity
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yuzhe Tang, Clinical Attending, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 42746034
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Marriage; Kidney Neoplasms; Surgery-Complications; Cohort Studies
Keywords: Marital Status; Kidney Cancer Surgery; Surgical Morbidity; Retrospective Cohort Study
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective cohort study

DETAILED DESCRIPTION:
Data source and study cohort:

We conducted a retrospective cohort study using the Premier Healthcare Database (PHD, Premier Inc., Charlotte, NC), an extensive, US hospital-based, all-payer database representing approximately 20% of annual United States inpatient discharges at community and academic centers. The International Classification of Diseases, ninth revision (ICD-9), and tenth revision (ICD-10) procedure codes were used to identify patients who had undergone elective kidney cancer surgery between the 15 years of study from 2003 to 2017. The cohort was then restricted based on appropriate ICD-9 and ICD-10 diagnosis codes to ensure that surgery was performed for a kidney mass. The study cohort was also limited to adult patients (age >= 18 years), "elective" cases based on administrative codes, as well as surgery on hospital day zero or one to minimize outlier patients who could skew the surgical outcomes.

Outcomes:

The primary outcome of this study was the 90-day complication rate. Complication rates were based on the Clavien-Dindo classification of surgical complications and divided into four categories: no complications, minor complications (Clavien grades 1, 2), and non-fatal major complications (Clavien grades 3, 4), and mortality (Clavien grade 5). Clinical systems also categorized complications (bleeding, cardiac, endocrine, gastrointestinal, infection, neurology, pulmonary, renal, soft tissue, urologic, venous thromboembolism) using Health Care Cost and Utilization Project Clinical Classification Software Level II or III designations; of note, the category for "surgical" complications was excluded given that all complications captured in this analysis are considered surgical complications. Secondary outcomes included patient disposition, length of hospital stay, and readmission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Surgery was performed for a kidney mass.
2. age >= 18 years
3. "elective" cases
4. Surgery was performed on the day0 or day1 after administration.

Exclusion Criteria:

1. ICD codes are not available.
2. Missing value of the primary outcomes and exposure.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study cohort was also limited to adult patients (age >= 18 years), "elective" cases based on administrative codes, as well as surgery on hospital day zero or one to minimize outlier patients who could skew the surgical outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 106752 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
surgical complications | 90 days after surgery
  Complication rates were based on the Clavien-Dindo classification of surgical complications and divided into four categories: no complications, minor complications (Clavien grades 1, 2), and non-fatal major complications (Clavien grades 3, 4), and mortality (Clavien grade 5).

SECONDARY OUTCOMES:
patient disposition | 90 days after surgery
  patient disposition was divided into home and none home such as skilled nursing or rehabilitation facility
readmission rates | 90 days after surgery
  readmission was defined as readmitted into the hospital for any reason

IPD SHARING:
Plan to Share IPD: Undecided